CLINICAL TRIAL: NCT01722383
Title: What Are the Determinations of Adult Progressive CKD? The Renal Impairment In Secondary Care (RIISC) Study
Acronym: RIISC
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Paul Cockwell, Consultant Nephrologist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK3917
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Urine, DNA, Saliva, Dental Plaque
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease: Stages 3-5 chronic kidney disease (pre-dialysis)

SUMMARY:
Chronic kidney disease (CKD) affects up to 16% of the adult population and is associated with significant morbidity and mortality. People at highest risk from progressive CKD are defined by a sustained decline in estimated glomerular filtration rate (eGFR) and/or the presence of significant albuminuria/proteinuria. Accurate mapping of the bio-clinical determinants of this group will enable improved risk stratification and direct the development of better targeted management for people with CKD. To address these requirements we have established the Renal Impairment in Secondary Care (RIISC) study; RIISC is enrolling a cohort of patients at high risk from progressive CKD and compiling a comprehensive and detailed bio-clinical phenotype, including vascular and oral health phenotyping, at enrolment and on subsequent follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Decline of eGFR of ≥5mls/min/year or ≥10mls/min/5years
* and/or urinary albumin-creatinine ration (ACR) ≥70 mg/mmol on three occasions
* and/or CKD 4 or 5 (pre-dialysis)

Exclusion Criteria:

* renal replacement therapy
* immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care kidney disease clinics
Sampling Method: Non-Probability Sample
Enrollment: 932 (Actual)
Dates: Start 2010-10; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants not alive | up to 10 years

SECONDARY OUTCOMES:
Number of participants who reach End Stage Kidney Disease | up to 10 years
  End Stage Kidney Disease describes a requirement for chronic dialysis treatment or a kidney transplant

OTHER OUTCOMES:
Number of participants who sustain one or more cardiovascular events | up to 10 years
Number of patients who require hospitalisation | up to 10 years
Number of patients who sustain a decline of kidney function | up to 10 years
  As measured by estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cockwell, MB BCh, Principal Investigator — University Hospital Birmingham
Locations (1):
- Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient data is being shared within the remit of the ethics for this study with collaborators

REFERENCES:
- [Derived] Sharma P, Fenton A, Dias IHK, Heaton B, Brown CLR, Sidhu A, Rahman M, Griffiths HR, Cockwell P, Ferro CJ, Chapple IL, Dietrich T. Oxidative stress links periodontal inflammation and renal function. J Clin Periodontol. 2021 Mar;48(3):357-367. doi: 10.1111/jcpe.13414. Epub 2021 Jan 28. PMID 33368493
- [Derived] Sharma P, Dietrich T, Sidhu A, Vithlani V, Rahman M, Stringer S, Jesky M, Kaur O, Ferro C, Cockwell P, Chapple IL. The periodontal health component of the Renal Impairment In Secondary Care (RIISC) cohort study: a description of the rationale, methodology and initial baseline results. J Clin Periodontol. 2014 Jul;41(7):653-61. doi: 10.1111/jcpe.12263. Epub 2014 May 14. PMID 24738870